CLINICAL TRIAL: NCT06719765
Title: The Correlation Between Forward Head Posture; Neck Pain, Neck Functional Ability and Deep Neck Core Strength in Jordanian University Students Having Chronic Non-specific Pain
Brief Title: The Correlation Between Forward Head Posture; Neck Pain, Neck Functional Ability and Deep Neck Core Strength in Jordan
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, Assistant professor kerolous ishak shehata, October 6 University
Other Study IDs: IRB#28\10\2024-2025
Record Dates: First submitted 2024-11-29; First posted 2024-12-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture
Keywords: forward head posture; neck pain; Jordanian university
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 60 Jordanian university students: Age range will between 18 to 25 years old
  - The study design will be observational cross sectional study

SUMMARY:
Is forward head posture correlated with neck pain, neck functional ability and deep neck core strength in Jordanian university students having chronic nonspecific pain.

DETAILED DESCRIPTION:
The study is an observational cross sectional study considering the effects of one of the most common spinal deformities such as forward head posture on the quality of life regarding Jordanian university students. University students are among the most common populations having these kinds of deformities because of using smart devices and studying for along periods of time in a faulty posture. 60 students "both male and females" having forward head posture with neck pain will be included in the study and different outcome measure as pain , functional ability and deep neck core strength will be measured to define the impact of this faulty posture on them. Pain measurement will be through using numeric rating scale for pain.

ELIGIBILITY:
Inclusion Criteria:

* The craniovertebral angle is less than 50 degrees .
* Age ranges from 18 to 25 years old
* Forward head is associated with neck pain.
* Studying hours more than 4 hours continuously per day

Exclusion Criteria:

* Previous surgery regarding the spine or shoulders.
* Vertebral fractures regarding the cervical spine or the skull.
* Positive neurological signs or evidence of spinal compression.
* headaches prior to the onset of neck pain and without cervical origin.
* Inner ear or vestibular Problems.

Ages: 18 Hours to 25 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will include 60 Jordanian university students (30 male & 30 female students)
  -Age range will between 18 to 25 years old
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Neck pain | 4 weeks
  Pain measurement will be through using numeric rating scale for pain which ranged from 0 means the least pain and 10 means the worst pain
Neck functional | 4 weeks
  Neck functional ability will be measured by neck disability index minimum score equal 10 (functional dependent) and maximum score equal 50 (functional independent)
Neck Core stability | 4 weeks
  Neck Core stability will be measured by pressure biofeedback unit
Craniovertebral angle | 4 weeks
  Craniovertebral angle will be measured by digital photography method

CONTACTS AND LOCATIONS:
Locations (1):
- AL-Zaytoonah University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No